CLINICAL TRIAL: NCT05491252
Title: A Patient-Centered Self-Management Intervention to Improve Glycemic Control, Self-Efficacy and Self-Care Behaviors in Adults With Type 2 Diabetes Mellitus: Randomized Controlled Trial
Brief Title: A Randomized Controlled Trial of Patient-Centered Self-Management Intervention in Adults With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shifa Tameer-e-Millat University (Other)
Responsible Party: Principal Investigator, Kainat Asmat, Kainat Asmat, Shifa Tameer-e-Millat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 335-21
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes, Self-management, Patient Centred Care, RCT
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: In parallel arm design, subjects are randomized to one or more study arms and each study arm will be allocated a different intervention. After randomization each subject stays in their assigned treatment arm for the duration of the study. Subjects receive the same treatment throughout the trial. The results are then compared.
Who Masked: Outcomes Assessor
Masking Description: Data Collectors / Outcome Assessors will be blinded of which treatment group subject is assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (CG) (No Intervention): The subjects in the Control Group (CG) will receive usual care as being received in study hospitals. Usual care at study hospitals involve consultaion with the physician which encompasses history taking, blood glucose measurement, prescription and provision of general education regarding lifestyle modification verbally or in the form of pamphelets.
- Intervention Group (IG) (Experimental): The subjects in the Intervention Group (IG) will receive usual care as well as a nurse-led PAtient CEntered Self-Management Intervention (PACE-SMI). PACE-SMI will be delivered for eight weeks duration comprising eight face to face individual and group educational, couselling and behavioral (ECB) training sessions in addition to telephonic reminders and a home visit by Principal Investigator (PI) and Research Assistants (RA). Outcome variables will be measured at three points in time (at baseline, at completion of intervention and lastly, after three months follow-up).
  Interventions: Behavioral: PAtient CEntered Self-Management Intervention (PACE-SMI)

INTERVENTIONS:
Behavioral: PAtient CEntered Self-Management Intervention (PACE-SMI) — Week 1: General disease knowledge. Week 2: Role of self-care behaviors towards effective management of type 2 diabetes, motivational video and real story of a diabetic patient to serve as a role-model. Lastly, provision of diabetes self-care guidebook.
  Week 3: Home visit to observe facilitators and barriers on initiating and maintaining behavioral change with social support as a key strategy.
  Week 4: ECB session on Diet. Week 5: ECB session on Physical Activity. Week 6: ECB session on Foot Care. Week 7: ECB session on Medication Adherence. Week 8: Booster session comprising reflection, performance feedback and review of behavioral goals fostering continued performance accomplishment and addressing difficulties of maintaining behaviour change over time.
  Arms: Intervention Group (IG)

SUMMARY:
Type 2 Diabetes Mellitus (DM) is a serious health problem for Pakistan and around the world due to its increasing prevalence and the risk of adverse health outcomes including kidney failure, heart attack, stroke, leg amputation and blindness. These problems reduce the quality of life of individuals with type 2 DM and increase their financial burden, thereby affecting the national economy. Given its huge health and economic impact, preventing type 2 DM progression and reducing the risk of associated complications requires immediate attention. Evidence suggests that self-management can slow the progression of type 2 DM, minimizes the risk of major complications and hence, lowers health-care costs. The purpose of this study is to test the effectiveness of a patient centered self-management intervention to improve health outcomes in adults with type 2 DM. It is expected that patients receiving this intervention would have improved health outcomes as compared to patients who did not.

DETAILED DESCRIPTION:
Background: In Pakistan, the rising burden of type 2 Diabetes Mellitus (DM) and its associated complications is considerably affecting the functional capacity of the individuals, their quality of life and demand for healthcare services with significant economic impact on health care system and the national economy. Given its enormous health and economic impact, preventing type 2 DM progression and reducing the risk of associated complications requires immediate attention. Evidence suggests that self-management can slow the progression of type 2 DM and minimize the risk of major complications thereby lowering health-care costs. Efective self-management on the other hand, demands patients' confidence and their full commitment to perform self care tasks necessitating a patient-centered approach.

Objective: To test the efficacy of a patient centered self-management intervention to improve glycemic control, self-efficacy and self-care behaviors in adults with type 2 DM.

Setting, Duration, Study Type: The study will be carried out as a randomized controlled trial (RCT) in four public tertiary care hospitals in Faisalabad, Pakistan.

Methods: A total 612 subjects will be recruited from out-patient departments (OPDs) of the study hospitals. Using random allocation 306 subjects will be assigned to the control group and 306 to the intervention group. Both the control group and the intervention group will receive usual care delivered at study hospitals. The intervention group will additionally receive a patient centered self-management Intervention for eight weeks duration.

Expected Outcome: If the study is able to show that the intervention group had improved glycemic control, self-efficacy and self-care behaviors than the control group. Then, employing hospital policies, this evidence-based care may be provided to all DM patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (aged 18 years or above)
2. Diagnosed with type 2 Diabetes Mellitus for at least 06 months duration.
3. Willing to participate in the study by signing of the consent form.

Exclusion Criteria:

1. Type 2 DM Patient with HbA1c < 7
2. Uncontrolled psychological comorbidity (psychosis, schizophrenia, dementia or severe learning difficulties).
3. Severe comorbidity that may limit participation (medical conditions such as cancer, stroke with disabilities, or need for regular dialysis etc. that preclude complete participation in this study).
4. Life expectancy of less than six months as determined by patient's primary physician.
5. Living outside of Faisalabad City.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Change in Glycemic Control (HbA1c) | HbA1c will be measured at three points in time (1) at baseline, (2) at completion of 8 weeks intervention, and (3) at three months follow-up
  HbA1c will be measured by collecting venous plasma samples and sending them to the single central laboratory to assure consistency and uniformity in methodology. The samples will be drawn by Data Collectors/Outcome Assessors and laboratory measurements will be performed by a trained laboratory technician.

SECONDARY OUTCOMES:
Self Efficacy | Self Efficacy will be measured at three points in time (1) at baseline, (2) at completion of 8 weeks intervention, and (3) at three months follow-up
  Self Efficacy will be measured on Diabetes management self-efficacy scale (DMSES). DMSES is a self-administered scale used to assess subjects's perceived confidence in their ability to manage blood sugar, diet, physical activity and foot care. The scale comprises of 20 items. Each item's response is rated on 11 point scale ranging from 'cant do at all (0)' to 'certain can do it' (10) with total score 0 to 200.
Self Care Behaviors | Self care behaviors will be measured at three points in time (1) at baseline, (2) at completion of 8 weeks intervention, and (3) at three months follow-up
  Self Care Behaviors will be measured on Summary of diabetes self-care activities (SDSCA). SDSCA is a self-reported scale to measure self-care activities across diverse components of diabetes self-management. SDSCA comprises of 25 items with each item measuring the frequency of self-care activities by asking how often several self-care activities were carried out over past seven days period. Each item's response is rated on 7 point scale ranging from '0' to '7' with total score ranging from 0 to 175. A higher score would be the frequency of performing self-care activities.

CONTACTS AND LOCATIONS:
Overall Officials: Khairunnisa Dhamani, PhD, Study Director — Shifa Tameer e Millat University, Islamabad, Pakistan; Erika Froelicher, PhD, Study Director — Shifa Tameer-e-Millat University; Raisa Gul, PhD, Study Director — Shifa Tameer-e-Millat University
Locations (4):
- Pakistan (4):
  - District Head Quarter (DHQ) Hospital, Faisalabad, Punjab Province
  - Allied Hospital, Faisalābad, Punjab Province
  - Government General Hospital, Faisalābad, Punjab Province
  - Punjab Social Security Hospital, Faisalābad, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Asmat K, Dhamani K, Froelicher ES, Gul R. A Patient-Centered Self-Management Intervention to Improve Glycemic Control, Self-Efficacy and Self-Care Behaviors in Adults with Type 2 Diabetes Mellitus: A SPIRIT Compliant Study Protocol for Randomized Controlled Trial. Diabetes Metab Syndr Obes. 2023 Jan 26;16:225-236. doi: 10.2147/DMSO.S385715. eCollection 2023. PMID 36760576